CLINICAL TRIAL: NCT00738374
Title: A Study of Chlorambucil Plus MabThera as Induction Therapy Followed in Responders by Maintenance Therapy Versus Observation on Response Rate in Patients >=60 Years With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study of MabThera (Rituximab) Plus Chlorambucil in Patients With Previously Untreated Chronic Lymphocytic Leukemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21445; 2008-001612-20
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Chlorambucil

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: chlorambucil

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 375mg/m2 iv on day 1 of course 3; 500mg/m2 iv on day 1 of courses 4-8 (induction phase); 375mg/m2 iv every 8 weeks (maintenance phase).
Drug: chlorambucil — 8mg/m2 po on days 1-7 of courses 1-8

SUMMARY:
This single arm study will assess the efficacy and safety of MabThera + chlorambucil as induction therapy, followed in responders by maintenance therapy or observation in elderly patients with previously untreated chronic lymphocytic leukemia. During the induction phase patients will receive 2 x 4 weekly courses of chlorambucil followed by 8 x 4 weekly courses of chlorambucil + MabThera. Subsequently, responders will be randomized to receive 12 doses of MabThera given every 8 weeks, or no further treatment. The anticipated time on study treatment is 2+ years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=60 years of age;
* CD20+ chronic lymphocytic leukemia (CLL);
* no previous treatment for CLL;
* ECOG performance status 0-1.

Exclusion Criteria:

* co-morbid conditions requiring long term use of systemic corticosteroids during study treatment;
* history of severe cardiac disease;
* transformation to aggressive B-cell malignancy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2008-11-03 (Actual); Primary Completion 2013-01-14 (Actual); Study Completion 2013-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (20):
- Italy (20):
  - Uni Degli Studi Di Bari, Policlinico; Cattedra Di Ematologia,Dipart. Di Medicina Interna E Publica, Bari, Apulia
  - Az. Osp. Pugliese; Dh Oncologico, Catanzaro, Calabria
  - P.O. Annunziata; U.O. Ematologia, Cosenza, Calabria
  - Ospedale Riuniti; Divisione Di Ematologia, Reggio Calabria, Calabria
  - Ospedale Cardarelli; Divisione Di Ematologia, Napoli, Campania
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - Arcispedale S. Anna; Sezione Di Ematologia, Ferrara, Emilia-Romagna
  - Ospedale S. Eugenio; Divisione Di Ematologia, Rome, Lazio
  - Universita' Degli Studi La Sapienza-Ist.Di Ematologia;Dip. Biotecnologie Cel CELLULARI ED EMATOLOGIA, Rome, Lazio
  - Uni Degli Studi Di Genova; 1A Divisione Di Ematologia, Genoa, Liguria
  - Ospedale Maggiore Di Milano; U.O. Ematologia I - Padiglione Marcora, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette;S.C. Ematologia, Turin, Piedmont
  - Ospedale Molinette - Universita' Di Torino; Cliniche Universitarie Ematologia I, Turin, Piedmont
  - Az. Osp. Papardo; Struttura Complessa Di Ematologia, Messina, Sicily
  - Ospedale Ferrarotto; Divisione Di Ematologia, Via S. Sofia 78, Sicily
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany
  - A.O. Universitaria Senese; Ematologia, Siena, Tuscany
  - Uni Degli Studi; Dip.Med.Clinica E Sperim. Ematologia, Padua, Veneto
  - Policlinico G. B. Rossi; Divisione Di Ematologia, Verona, Veneto

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorambucil (CLB) Plus (+) Rituximab (R): Induction Treatment: Participants completed an 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 milligrams per square meter (mg/m^2), orally (PO) as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, intravenously (IV), on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8. Participants with complete response (CR), complete response with incomplete bone marrow recovery (CRi), or partial response (PR) were randomized to receive either rituximab, 375 mg/m^2, IV, every 8 weeks for up to 24 months, or to be observed for up to 24 months with no further treatment.
- CLB + R: Completed Induction Treament But Not Randomized: Participants completed an 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 mg/m^2, PO as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, IV, on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8. Participants were not randomized to receive further treatment or observation.
- CLB + R: Maintenance Treatment: Participants completed an 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 mg/m^2, PO as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, IV, on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8. Participants with CR, CRi, or PR were randomized to receive rituximab, 375 mg/m^2, IV, once every 8 weeks for a total of 12 infusions for up to 24 months.
- CLB + R: Observation: Participants completed an 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 mg/m^2, PO as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, IV, on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8. Participants with CR, CRi, or PR were randomized to be observed for up to 24 months and received no further treatment.
Period: Induction Treatment Phase
Arm/Group | Chlorambucil (CLB) Plus (+) Rituximab (R): Induction Treatment | CLB + R: Completed Induction Treament But Not Randomized | CLB + R: Maintenance Treatment | CLB + R: Observation
Started | 97 | 0 | 0 (Participants were randomized at the end of the Induction Treatment Phase.) | 0 (Participants were randomized at the end of the Induction Treatment Phase.)
Completed | 73 | 0 | 0 | 0
Not Completed | 24 | 0 | 0 | 0
Not completed — Adverse Event | 14 | 0 | 0 | 0
Not completed — Disease progression/relapse/stable | 4 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Maintenance Treatment/Observation Phase
Arm/Group | Chlorambucil (CLB) Plus (+) Rituximab (R): Induction Treatment | CLB + R: Completed Induction Treament But Not Randomized | CLB + R: Maintenance Treatment | CLB + R: Observation
Started | 0 (Participants were randomized to either maintenance therapy or observation at the end of induction.) | 7 | 34 | 32
Completed | 0 | 0 | 27 | 20
Not Completed | 0 | 7 | 7 | 12
Not completed — Adverse Event | 0 | 1 | 2 | 0
Not completed — Disease progression/relapse/stable | 0 | 4 | 5 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- CLB + R: Not Randomized: Participants began a 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 mg/m^2, PO as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, IV, on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8. Participants who completed the induction treatment with CR, CRi, or PR were randomized to receive either rituximab, 375 mg/m^2, IV, every 8 weeks for up to 24 months, or to be observed for up to 24 months with no further treatment.
- Total: Total of all reporting groups
Arm/Group | CLB + R: Not Randomized | CLB + R: Maintenance Treatment | CLB + R: Observation | Total
Number analyzed (Participants) | 31 | 34 | 32 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (6.5) | 69.8 (5.4) | 70.2 (5.1) | 71.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 9 | 32
  Male | 18 | 24 | 23 | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Documented CR, CRi, or PR at the End of Induction Treatment
Description: CR defined as: 1) laboratory CR: peripheral blood lymphocytes (PBL) less than (<) 4000/microliter (μL), neutrophils (PMN) greater than (>) 1500/μL, platelets >100,000/μL, and hemoglobin (Hb) >11 grams per deciliter (g/dL); 2) clinical CR: lymph nodes (LN) <1.5 centimeter (cm), and no constitutional symptoms, hepatomegaly (HM) or splenomegaly (SM); 3) instrumental CR: LN <1.5 cm and no HM/SM, and 4) bone marrow (BM) CR: normocellular aspirate/biopsy for participant age <30 percent (%) lymphocytes, and no B cell lymphoid nodules. CRi was defined as CR with anemia, thrombocytopenia, or neutropenia not related to chronic lymphocytic leukemia (CLL), with no clonal infiltrate in aspirate or biopsy. PR defined as: a 50% decrease in PBL, a 50% decrease in LN size, no increase in LN size, no new enlarged LN, a 50% reduction from baseline (BL) in the HM/SM, and 1 of the following: PMN >1500/μL, platelets >100,000/μL or >50% improvement from BL, and Hb >11.0 g/dL or >50% improvement from BL.
Time Frame: Month 10
Population: Intent to treat (ITT) population: all consented participants who received at least 1 dose of rituximab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CLB + R: All Participants: Participants completed an 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 mg/m^2, PO as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, IV, on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8. Participants with CR, CRi, or PR were randomized to receive either rituximab, 375 mg/m^2, IV, once every 8 weeks for up to 24 months (up to 12 infusions), or to be observed for up to 24 months with no further treatment.
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
percentage of participants | 82.4 [74.25 to 90.46]
Statistical Analysis 1: Comparison: CLB + R: All Participants; Analysis compared responders and non-responders; Test type: Superiority or Other; p = 0.0008, Chi-squared

2. Secondary Outcome: Percentage of Participants With Documented CR, CRi, or PR at the End of Study
Description: CR defined as: 1) laboratory CR: PBL <4000/μL, PMN > 1500/μL, platelets > 100,000/μL, and Hb > 11 g/dL; 2) clinical CR: LN < 1.5 cm, and no constitutional symptoms, HM or SM; 3) instrumental CR: LN < 1.5 cm and no HM/SM, and 4) bone marrow CR: normocellular aspirate/biopsy for participant age < 30% lymphocytes, and no B cell lymphoid nodules. CRi was defined as CR with anemia, thrombocytopenia, or neutropenia not related to CLL, with no clonal infiltrate in aspirate or biopsy. PR defined as: a 50% decrease in PBL, a 50% decrease in LN size, no increase in LN size, no new enlarged LN, a 50% reduction from BL in the HM/SM, and 1 of the following: PMN > 1500/μL, platelets > 100,000/μL or > 50% improvement from BL, and Hb >11.0 g/dL or > 50% improvement from BL.
Time Frame: Month 35
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLB + R: Maintenance Treatment | CLB + R: Observation
Number analyzed (Participants) | 34 | 32
percentage of participants | 55.9 [39.19 to 72.57] | 34.4 [17.92 to 50.83]
Statistical Analysis 1: Comparison: CLB + R: Maintenance Treatment vs CLB + R: Observation; Test type: Superiority or Other; p = 0.0795, Chi-squared

3. Secondary Outcome: Percentage of Participants With CR, CRi, PR, Stable Disease (SD), Progressive Disease (PD), Relapse, or Nodular PR at the End of Induction Treatment
Description: CR, CRi, and PR as previously defined. PD was defined by 1 of the following: 1) lymphadenopathy: any new lesion, HM/SM, or other organ infiltrates, or a greater than or equal to (≥) 50% increase in greatest diameter of any previously noted lesion; 2) a ≥ 50% increase in previously noted HM/SM, or new appearance of HM/SM; 3) a ≥ 50% increase in blood lymphocyte count with at least 5000 B lymphocytes/μL; 4) transformation to a more aggressive histology, e.g., Richter's syndrome; or 5) occurrence of cytopenia attributable to CLL. SD was defined by the absence of necessary criteria to achieve CR or PR, but no advancement to PD. Relapse was defined by a previously noted CR or PR with advancement to PD after a period of ≥ 6 months. Nodular PR was defined by the presence of residual lymphoid nodules.
Time Frame: Month 10
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- CLB + R: Induction Treatment: Participants completed an 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 mg/m^2, PO as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, IV, on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8.
Arm/Group | CLB + R: Induction Treatment
Number analyzed (Participants) | 85
percentage of participants
  CR | 16.5
  CRi | 2.4
  PR | 60.0
  SD | 4.7
  PD | 3.5
  Relapse | 0.0
  Nodular PR | 3.5
  Unknown | 9.4

4. Secondary Outcome: Percentage of Participants With CR, PR, SD, PD, Relapse, or Nodular PR at the End of Study
Description: CR, and PR as previously defined. PD was defined by 1 of the following: 1) lymphadenopathy: any new lesion, HM/SM, or other organ infiltrates, or a ≥ 50% increase in greatest diameter of any previously noted lesion; 2) a ≥50% increase in previously noted HM/SM, or new appearance of HM/SM; 3) a ≥50% increase in blood lymphocyte count with at least 5000 B lymphocytes/μL; 4) transformation to a more aggressive histology, e.g., Richter's syndrome; or 5) occurrence of cytopenia attributable to CLL. SD was defined by the absence of necessary criteria to achieve CR or PR, but no advancement to PD. Relapse was defined by a previously noted CR or PR with advancement to PD after a period of ≥6 months. Nodular PR was defined by the presence of residual lymphoid nodules.
Time Frame: Month 35
Population: All randomized participants who were assessed at Month 35 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CLB + R: Maintenance Treatment | CLB + R: Observation
Number analyzed (Participants) | 31 | 28
percentage of participants
  CR | 32.3 | 21.4
  PR | 29.0 | 14.3
  SD | 3.2 | 7.1
  PD | 29.0 | 39.3
  Relapse | 6.5 | 14.3
  Nodular PR | 0.0 | 3.6

5. Secondary Outcome: Number of Participants With Immunophenotypic CR - BM, Immunophenotypic CR - Peripheral Blood (PB), Molecular CR - BM, or Molecular CR - PB at the End of Induction Treatment
Description: Immunophenotypic CR was defined as the absence of minimal residual disease (MRD) evaluated in participants with CR by 4-color flow cytometry of PB and BM B cells to confirm that tissue was comprised of non-CLL cells. Molecular CR was defined as the absence of MRD evaluated in participants with CR by quantitative polymerase chain reaction (PCR) in PB and BM B cells to confirm that tissue was comprised of non-CLL cells.
Time Frame: Month 10
Population: ITT population
Measure: Number; unit: participants
Arm/Group | CLB + R: Induction Treatment
Number analyzed (Participants) | 85
participants
  Immunophenotypic CR - BM | 2
  Immunophenotypic CR - PB | 3
  Molecular CR - BM | 0
  Molecular CR - PB | 0

6. Secondary Outcome: Percentage of Participants With CR, CRi, PR, SD, PD, or Relapse at the End of Study
Description: CR, CRi, PR, SD, PD, relapse, and nodular PR as previously defined.
Time Frame: Month 35
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | CLB + R: Maintenance Treatment | CLB + R: Observation
Number analyzed (Participants) | 34 | 32
percentage of participants
  CR | 29.4 | 18.7
  CRi | 0.0 | 0.0
  PR | 26.4 | 12.5

7. Secondary Outcome: Percentage of Participants With Immunophenotypic CR - BM or Immunophenotypic CR - PB at the End of Study
Description: Immunophenotypic CR was defined as the absence of MRD evaluated in participants who achieved CR by 4-color flow cytometry of PB and BM B cells to confirm that tissue was comprised of non-CLL cells.
Time Frame: Month 35
Population: All randomized participants, only participants with a confirmed CR were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CLB + R: Maintenance Treatment
Number analyzed (Participants) | 10
percentage of participants
  Immunophenotypic CR - BM | 10.0
  Immunophenotypic CR - PB | 30.0

8. Secondary Outcome: Percentage of Participants With Molecular CR - BM or Molecular CR - PB at the End of Study
Description: Molecular CR was defined as the absence of MRD evaluated in participants who achieved CR by quantitative PCR in PB and BM B cells to confirm that tissue was comprised of non-CLL cells.
Time Frame: Month 35
Population: All randomized participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | CLB + R: Maintenance Treatment
Number analyzed (Participants) | 3
percentage of participants
  Molecular CR - BM | 100.0
  Molecular CR - PB | 33.3

9. Secondary Outcome: Number of Participants With Disease Progression, Relapse, Death, Withdrawal Because of an Adverse Event (AE), or New CLL Treatment
Description: Event-free Survival (EFS) was defined as the time from the first dose of study treatment to the date of first documentation of disease progression, relapse for participants with previous CR, death due to any cause, withdrawal due to AE, or beginning new CLL treatment. CR and PD as previously defined. Participants were censored at the time of data cut-off to the most recent date of disease assessment. Participants without a post-BL disease assessment were censored at the time of first dose of study treatment.
Time Frame: Screening, Days 1 and 15 of Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
participants | 43

10. Secondary Outcome: EFS
Description: The median time, in days, from the the date of first dose of study treatment to the date of first documentation of disease progression, relapse for participants with CR, death due to any cause, withdrawal due to AE, or new CLL treatment. CR and PD as previously defined. Participants were censored at the time of data cut-off to the most recent date of disease assessment. Participants without a post-BL disease assessment were censored at the time of first dose if study treatment. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: as for outcome 9
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
days | 1051 [768 to 1164]

11. Secondary Outcome: Number of Participants With Disease Progression or Death
Description: Progression-free survival (PFS) was defined as the time from the first dose of study treatment to the first documentation of disease progression or death. PD as previously defined. Participants who were withdrawn from the study without documented disease progression were censored at the date of the last tumor assessment when the participant was known to be progression-free. Participants without a post-BL tumor assessment, but known to be alive, were censored at the time of the first dose of study treatment.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
participants | 35

12. Secondary Outcome: PFS
Description: The median time, in days, from the date of the first dose of study treatment to the date of first documentation of disease progression or death. CR and PD as previously defined. Participants who were withdrawn from the study without documented disease progression were censored at the date of the last tumor assessment when the participant was known to be progression-free. Participants without a post-BL tumor assessment, but known to be alive, were censored at the time of the first dose of study treatment. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
days | 1059 [1010 to 1205]

13. Secondary Outcome: Number of Participants With New CLL Treatment or Death
Description: Time to new CLL treatment (TTNT) was defined as the time from the first dose of study treatment to the date of new CLL treatment received or the date of death from any cause. Participants who did not receive new CLL treatment and were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without a follow-up assessment were censored at the day of last dose of study treatment.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
participants | 22

14. Secondary Outcome: Time to Next Treatment (TTNT)
Description: The mean time, in days, from the date of the first dose of study treatment to the date of new CLL treatment or the date of death from any cause. Participants who did not receive new CLL treatment and were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without a follow-up assessment were censored at the day of last dose of study treatment. Mean survival time and it's standard error (SE) were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: ITT population
Measure: Mean (Standard Error); unit: days
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
days | 1048.19 (31.86)

15. Secondary Outcome: Number of Participants Who Died
Description: Overall Survival (OS) was defined as the time from the date of the first dose of study treatment to the date of death due to any cause. Participants were censored at the date of the last follow-up assessment. Participants without a follow-up assessment were censored at the day of last dose of study treatment.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
participants | 8

16. Secondary Outcome: OS
Description: The mean time, in days, from the date of the first dose of study treatment to the date of death due to any cause. Participants were censored at the date of the last follow-up assessment. Participants without a follow-up assessment were censored at the day of last dose of study treatment. The mean survival time and it's SE were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: ITT population
Measure: Mean (Standard Error); unit: days
Arm/Group | CLB + R: All Participants
Number analyzed (Participants) | 85
days | 1135.04 (24.25)

17. Secondary Outcome: Number of Participants With PD or Death After a Confirmed CR, CRi, or PR
Description: Duration of response was defined as the time from the date of the first documented CR, CRi, or PR to the date of disease progression or death. CR, CRi, PR, and PD as previously defined. Participants with no documented PD after CR, CRi, or PR were censored at the last date at which they were known to have had CR, CRi, or PR, respectively.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | CLB + R: Maintenance Treatment | CLB + R: Observation
Number analyzed (Participants) | 34 | 32
participants | 11 | 15

18. Secondary Outcome: Duration of Response
Description: The mean time, in days, from the date of first documented CR, CRi or PR to the date disease progression or death. CR, CRi, PR, and PD as previously defined. Participants with no documented PD after CR, CRi, or PR were censored at the last date at which they were known to have had CR, CRi, or PR, respectively.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: All randomized participants.
Measure: Mean (Standard Error); unit: days
Arm/Group | CLB + R: Maintenance Treatment | CLB + R: Observation
Number analyzed (Participants) | 34 | 32
days | 840.87 (29.71) | 747.82 (55.77)
Statistical Analysis 1: Comparison: CLB + R: Maintenance Treatment vs CLB + R: Observation; Test type: Superiority or Other; p = 0.2712, Log Rank

19. Secondary Outcome: Number of Participants With PD or Death After a Confirmed CR/CRi
Description: Disease-free survival was defined at the time from the date of first documented CR or CRi to the date of disease progression or death. CR, CRi, and PD as previously defined. Participants with no documented PD after CR or CRi were censored on the last date at which they were known to have had CR or CRi.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: All randomized participants with a confirmed CR or CRi were included in the analysis.
Measure: Number; unit: participants
Arm/Group | CLB + R: Maintenance Treatment | CLB + R: Observation
Number analyzed (Participants) | 16 | 15
participants | 2 | 8

20. Secondary Outcome: Disease-Free Survival
Description: The mean time, in days, from the date of first documented CR or CRi to the date of disease progression or death. CR, CRi, and PD as previously defined. Participants with no documented PD after CR or CRi were censored on the last date at which they were known to have had CR or CRi. In both groups, the mean survival time and its standard error were underestimated because the largest observation was censored and the estimation was restricted to the largest event time.
Time Frame: Screening, Day 1 Courses 1-8 (4-week courses) and Day 1 of Courses 10-35 (4-week courses) for up to 35 months.
Population: All randomized participants.
Measure: Mean (Standard Error); unit: days
Arm/Group | CLB + R: Maintenance Treatment | CLB + R: Observation
Number analyzed (Participants) | 34 | 32
days | 699.91 (68.89) | 732.28 (63.37)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from Screening through the Final Visit or withdrawal from study, approximately 35 months.
Description: All participants who received at least 1 dose of chlorambucil or rituximab were included in the analysis.
Groups:
- CLB + R: Induction Treatment: Participants completed an 8-month induction treatment phase where they received 8 (4-week) courses of treatment consisting of: CLB, 8 mg/m^2, PO as film-coated tablets, daily (dose could be divided in halves or thirds to prevent nausea), on Days 1-7 of Courses 1 and 2, Days 2-8 of Course 3, and Days 1-7 of Courses 4-8; and rituximab, 375 mg/m^2, IV, on Day 1 of Course 3, and 500 mg/m^2, IV, on Day 1 of Courses 4-8. Participants with CR, CRi, or PR were randomized to receive either rituximab, 375 mg/m^2, IV, once every 8 weeks for up to 24 months (up to 12 infusions), or to be observed for up to 24 months with no further treatment.
Arm/Group | CLB + R: Induction Treatment | CLB + R: Maintenance Treatment | CLB + R: Observation
Serious Adverse Events (participants affected / at risk) | 17/97 | 4/34 | 4/32
Other Adverse Events (participants affected / at risk) | 73/97 | 25/34 | 17/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLB + R: Induction Treatment (N=97) | CLB + R: Maintenance Treatment (N=34) | CLB + R: Observation (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Herpes zoster oticus (Infections and infestations) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mixed oligo-astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Porocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLB + R: Induction Treatment (N=97) | CLB + R: Maintenance Treatment (N=34) | CLB + R: Observation (N=32)
Anaemia (Blood and lymphatic system disorders) | 14 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 5 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 31 | 5 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 1 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 0
Dyskinesia oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 0 | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0
Asthenia (General disorders) | 4 | 1 | 0
Chest pain (General disorders) | 3 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 5 | 0 | 3
Hyperpyrexia (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 3 | 0 | 1
Infusion related reaction (General disorders) | 6 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 2 | 0
Pyrexia (General disorders) | 11 | 0 | 2
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Multiple allergies (Immune system disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 2 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 3 | 0 | 1
Herpes zoster oticus (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 1
Productive cough (Infections and infestations) | 1 | 0 | 0
Pyrexia (Infections and infestations) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 2 | 1
Hypotension (Vascular disorders) | 3 | 0 | 0
Thyroid disorder (Endocrine disorders) | 0 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Tongue dry (Gastrointestinal disorders) | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 4 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine increased (Investigations) | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0
Peyronie's disease (Reproductive system and breast disorders) | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 0 | 0 | 1
Knee operation (Surgical and medical procedures) | 0 | 0 | 1
Carotid artery stenosis (Vascular disorders) | 0 | 1 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.